Risk of revision and other complications following knee arthroplasty in patients previously exposed to bariatric surgeries: A nationwide, register-based study

#### Authors/Collaborators:

Saber M. Saber<sup>1,2,4</sup>, MD, PhD Fellow; Janne Petersen MSc, PhD, Associate Professor<sup>3,6</sup>; Robin Christensen<sup>2,5</sup>, MSc, PhD, Professor; Espen Solem, MD, PhD, Associate Professor<sup>3,4</sup>; Søren Overgaard, MD, DmSci, Professor<sup>1,4</sup>

#### Affiliations:

1. Department of Orthopaedic Surgery and Traumatology, Copenhagen University Hospital, Bispebjerg and Frederiksberg, Copenhagen, Denmark; 2. Section for Biostatistics and Evidence-Based Research, the Parker Institute, Copenhagen University Hospital, Bispebjerg and Frederiksberg, Copenhagen, Denmark; 3. Copenhagen Phase IV unit (Phase4CPH), Department of Clinical Pharmacology and Center of Clinical Research and Prevention at Copenhagen University Hospital, Bispebjerg and Frederiksberg; 4. University of Copenhagen, Department of Clinical Medicine, Faculty of Health and Medical Sciences; 5. Research Unit of Rheumatology, Department of Clinical Research, University of Southern Denmark, Odense University Hospital, Denmark & 6. Section of Biostatistics, Department of Public Health, University of Copenhagen, Copenhagen, Denmark.

**Abstract** 

Background: Previous studies have investigated the outcomes of Knee Arthroplasty (KA) following Bariatric

Surgery (BAS), but with substantial limitations as not stratifying for Body Mass Index (BMI) at time of KA or

not addressing the type of BAS (gastric bypass, banding or sleeve). Since BMI varies greatly in patients with

previous BAS, it is likely that BMI affects outcomes after KA in BAS-operated patients.

Objective: Based on the Danish national registers and databases. The objective of this study is to analyse

the association between exposure to BAS prior to KA and the following outcomes: 1) the risk of revision, 2)

use of antibiotics and 3) mortality. Furthermore, we want to test whether the association is modified by BMI

status at the time KA surgery (i.e., non-obese, obese and morbidly obese patients).

Methods/Design: The study is a nationwide, register-based cohort study. The study will follow the

reporting of studies conducted using observational routinely-collected data statement for

PharmacoEpidemiology (RECORD-PE) guidelines. We will compare the risk of revision after primary KA

between patients with or without prior BAS. We will stratify the for BMI (non-obese: BMI < 30 kg/m2, obese:

BMI 30-39 kg/m2, morbidly obese: BMI ≥ 40 kg/m2) at time of KA and the type of KA (i.e., Total Knee

Arthroplasty (TKA) or Unicondylar Knee Arthroplasty (UKA)).

Exposures and outcomes: Exposure will be defined as BAS prior to KA. Outcomes are 1) revision due to all

causes; 2) revision due to infection; 3) Knee related use of antibiotics within 30- and 90 days after the index

KA; 4) Antibiotic use due to other causes within 30- and 90 days after the index KA and 5) mortality rate

within 2 years following the index KA. We will use BMI, year of KA, year of BAS, sex, household income,

highest completed education, comedication, Elixhauser Comorbidity Measure (ECM) and the NOMESCO

(Nordic Medico-Statistical Committee) Classification of Surgical Procedures for stratifying and matching...

Multiple sensitivity analyses will be performed to investigate the influence of time between BAS and KA;

and the type of BAS on the outcomes.

**Perspectives**: The purpose of this study is to estimate the risk of complications following KA in patients with

previous exposure to BAS and it is anticipated that findings from this study would potentially help shared-

decision making between the surgeon and patient - weighing the risks and benefits and by that, optimise

selection of the right patients.

Keywords: Knee Arthroplasty, Bariatric Surgery, Risk of Revision, Register, Osteoarthritis

## **INTRODUCTION**

Knee Arthroplasty (KA) have been estimated to have a 15-years survival rate of around 93%.¹ The main indications for revision after knee arthroplasty are aseptic loosening, infection and pain.² Surgical risk factors for revision include uncemented components, implant malalignment and longer length of operation. Patient-related risk factors include obesity, male sex and younger age at time of KA.³-8 Obese patients (BMI>30 kg/m²) have a higher risk for revision, deep and superficial infection, wound dehiscence and readmission following KA.⁵ As obesity is a major risk factor much attention has been paid to weight loss before surgery. bariatric surgery (BAS) is an efficient weight-reducing intervention and can lead to a decrease in excess weight by up to 74% through all types of bariatric surgeries.³ The prevalence of BAS-operated patients is increasing due to the increased obesity worldwide.¹o Whether BAS previous to KA is advantageous is disputed, mainly because BAS carries possible long-term complications, which vary depending on the type of BAS.¹¹¹₁¹² For example, late, non-surgical complications such as nutritional deficiencies of micronutrients and vitamins (including vitamin D) may impact bone metabolism and immune capacity and hence increase the risk of revision after KA, despite the weight loss achieved by BAS.³³

Previous studies have investigated the outcomes of KA after BAS, but with substantial limitations. <sup>14,-24</sup> A recent RCT concluded a reduced risk of complications after KA in patients exposed to BAS. The trial was underpowered (and prematurely terminated) for important outcomes and has limited external validity due to unclear exclusion criteria and a high number of excluded patients. <sup>16</sup> Other limitation is the treatment of BAS as a homogenous group without stratifying for BMI at time of KA or type of BAS (gastric bypass, banding or sleeve). <sup>17,-24</sup> For instance, various studies have reported that the Body Mass Index (BMI) of the BAS-groups at the time of knee arthroscopy (KA) falls within a broad range of 23-57 kg/m2. <sup>21,22,24</sup> This significant variance in BMI suggests considerable heterogeneity within this group. Furthermore, this wide range in BMI could potentially influence the outcomes reported in these studies. Moreover, some researchers did not report the registered body mass index (BMI) at the time of KA. Instead, they relied on ICD-9 codes for their data. <sup>17-20,23</sup> This approach results in a comparison between two groups that are fundamentally dissimilar. This is because ICD-9 codes do not accurately reflect overweight conditions, and in a US sample, only 15.1% of overweight patients were assigned relevant ICD-9 codes. <sup>25</sup>

## Objective

The objective of this study is to analyse the association between exposure to BAS prior to KA and the following outcomes: 1) the risk of revision, 2) use of antibiotics and 3) mortality. Furthermore, we want to test whether the association is modified by BMI at the time KA surgery (i.e., non-obese, obese and morbidly

obese patients). This would help the surgeon in weighing the risks and benefits and by that, selecting the right patient for operation.

#### **METHODS**

### Study design

The study is a nationwide, register-based cohort study. The study will be reported following the REporting of studies Conducted using Observational Routinely-collected Data statement for PharmacoEpidemiology (RECORD-PE) guidelines. <sup>26</sup> We will compare the risk of revision after primary KA in the period from 2011 and 2 years earlier to data-extraction date stratified for exposure to BAS prior to their KA. We will further stratify for BMI (non-obese: BMI < 30 kg/m², obese: BMI 30-39 kg/m², and morbidly obese: BMI  $\geq$  40 kg/m²) at time of KA and the type of KA (i.e., Total Knee Arthroplasty (TKA) or Unicondylar Knee Arthroplasty (UKA)).

## Setting

There are approximately 5.8 million inhabitants in Denmark, and every citizen has a unique 10-digit Civil Personal Register (CPR) number in the Danish Civil Registration System (DCRS), and by this number citizens can be cross-linked across different databases and be traced until death or immigration.

#### **Data sources**

The Danish Civil Registration System (DCRS) contains information on the CPR number, vital and migrant status, cohabiting status, and municipality of residence.<sup>27</sup>

The Danish Knee Arthroplasty Register (DKR) is nation-wide register that contains information on all primary knee arthroplasty procedures and revisions performed in Denmark, e.g., baseline characteristics as age, sex, BMI, at the time of KA operation. The registry started in 1997 and the reporting to the registry became mandatory since 2006. DKR is known for high degree of coverage and completeness.<sup>28,29</sup>

The Danish Microbiology Database (MiBa) is a national database containing data from all samples received by the Danish clinical microbiology departments from both hospitals and general practices with complete coverage since 2010. <sup>30</sup>

The Danish National Patient Register (DNPR) is a valuable tool for epidemiological research, providing longitudinal registration of diagnoses, treatments, and examinations derived from every hospital contact in Denmark with complete nationwide coverage since 1978. <sup>31</sup>

The Danish National Prescription Registry has kept information on all prescriptions for drugs dispensed by community pharmacies in Denmark since 1994 according to Anatomical Therapeutic Chemical (ATC) classification system (ATC codes). Data from the Danish National Prescription Registry does not include hospital dispensaries.<sup>32</sup>

The Danish Registers on Personal Income and Transfer Payments contains more than 160 variables including salaries, entrepreneurial income, taxes, public transfer payments, capital income, private pension contributions, and pay-outs. In addition, Statistics Denmark provide more detailed registers on specific income transfers, including sickness benefit, old age pension, disability pension, and cash and unemployment benefits.<sup>33</sup>

The Danish Population Education Register provides information on education status on Danish population, and it carries high degree of validity and coverage.<sup>34</sup>

## Study population

We will include patients with primary/idiopathic or secondary (due to meniscus or cruciate ligament lesion) osteoarthritis (OA) who received primary KA in the period from 2011 and 2021. Patients will be identified from the DKR. Patients are followed for 2 years, until first revision, death or migration, whichever comes first.

#### **Variables**

#### **Outcomes:**

- 1. Revision due to any cause at two different observation periods within 1) 90 days and b) 2 years following KA. Revision surgery with debridement and/or exchange of at least one component will be based on a composite endpoint (34)
- 2. Revision due to infection within 1) 90 days and b) 2 years following KA: our definition of infection is adapted from the European Bone and Joint Infection Society (EBJIS) criteria <sup>35</sup> as at least one of the following
  - A. DKR-registered revision surgery due to infection.
  - B. At least 2 deep-tissue samples of phenotypically indistinguishable bacteria isolated from at least 3 deep-tissue samples
  - C. One or more positive intraoperative samples from a closed fluid aspirate AND a biopsy (fluid AND tissue) of phenotypically indistinguishable bacteria isolated.
- 3. Antibiotic use within 30- and 90-days following KA as measure of knee related infection will be defined as the use of one of the following oral antibiotics: dicloxacillin, flucloxacillin,

phenoxymethylpenicillin, or amoxicillin as suggested by Milandt et al.<sup>36</sup> Other antibiotics recommended by the international consensus for treating joint infections will also be considered knee-related: oral ciprofloxacin, roxithromycin, linezolid, cefuroxime and cefalexin. <sup>37</sup>

- 4. Antibiotic use within 30- and 90-days following KA due to other causes: any oral antibiotic other than the forementioned ones.
- 5. Mortality registered in the DCRS by date up to 2 years following KA surgery.

#### Covariates

We will identify our cohort as patients, who had a BAS before the date of index arthroplasty based on the NOMESCO (Nordic Medico-Statistical Committee) Classification of Surgical Procedures from the DNPR (KJDF10 & KJDF11 [gastric bypass]; KJDF20 & KJDF21 [gastric banding]; KJDF40, KJDF41, KJDF96 & KJDF97 [gastric sleeve]). The comparator (unexposed) group will be patients without BAS before KA.

BMI category and the type of KA (TKA and UKA). will be used for stratifying into subgroups, differentiating individuals into appropriate baseline strata. For matching we will be using the following pre-KA-exposure covariates: age (years) at the year of KA, sex (male/female), household income (at the year of KA, categorized into quartiles), highest completed education (at the year of KA, categorized into 3 categories: <11, 11 to 15, and >15 years).

Comedication (at least one redeemed prescription 365 days earlier to index KA - 60 days for antibiotics): 1) Glucose-lowering due to the association between DM and surgical complications.  $^{38,39}$  2) Antithrombotic medications and 3) NSAIDs because of the possible postoperative bleeding-related complications  $^{40}$  and 4) Antiresorptives due to the possible increased risk of revision.  $^{41}$  The last covariate to be included in matching and adjustment is Elixhauser Comorbidity Measure (ECM) (at the year of KA, categorized into 3: 0, 1-2 and  $\geq$  3), ECM is validated comorbidity scoring measure that has shown highest discriminative ability for the occurrence of all categories of postoperative adverse outcomes following orthopedic surgeries.  $^{42-44}$ 

For sensitivity analyses we will analyse the type of BAS and the calendar year of BAS and the calendar year of KA.

## Database construction and handling

We will extract data from all patients receiving KA in period from 2011 and 2023 the DKR, the dataset will be enriched with the relevant variables by cross-linking the CPR numbers from the MiBa and will be sent to

Statistics Denmark, where the baseline socioeconomic data will be supplied. The database will be then enriche with baseline health-related data from the Danish Health Data Authority (DHDA). The final database will be kept and handled inside an encrypted server belonging to Statistics denmark. Data is handled in the most recent version of R (www.r-project.org). The primary author (SMS) will be responsible for data management.

## Data control and editing

In case of bilateral KA, the first one will be treated as study unit. In case of simultaneous bilateral KA, patients will be excluded.

We expect some missing values in our study and these values will be omitted, no data imputation will be used.

Extreme values for continuous variables will be tested by using plots and histograms to identify the possible entry-errors.

In case of abnormal data entries, e.g., wrong date format, it will be corrected if possible, otherwise the values will be omitted.

#### Statistical Methods

We will use descriptive statistics for the baseline characteristics of the two groups stratified for BMI and the type of KA. To address possible survival bias, number of deaths in the exposed and non-exposed groups will be reported.

First, we will run a non-adjusted (crude) analysis comparing outcomes between patients exposed and unexposed to BAS. Then we will perform a propensity score matched analysis, where we do exact matching based on BMI (non-obese: BMI < 30 kg/m², obese: BMI 30-39 kg/m², morbidly obese: BMI ≥ 40 kg/m²) and the type of KA (i.e., TKA or UKA). Propensity scores will be estimated using a logistic regression model and will be based the forementioned covariates. We will use greedy match algorithm in a ratio of up to 1:5 of patients exposed to bariatric surgery and those who are not, in order to minimize the mean squared error of the estimated treatment effect in several scenarios, difference of maximum of 0.2 logit will be used in propensity score matching <sup>45</sup>. Following that, we will do a propensity score matched analysis with interaction term for BMI.

For dichotomous outcomes, a cox regression will be performed to report hazards ratio with the corresponding two-sided 95% confidence intervals (Cis) and a p-value of <0.05 will be considered as statistically significant.

To validate the propensity score matching, we will report the standardized differences of the means (or medians) of continuous variables or the prevalence of dichotomous baseline covariates between each set of groups by using the standardised differences. We will apply a standardized difference of  $\geq 0.25$  to indicate that there might be a meaningful imbalance in the baseline covariate.

# Sensitivity analyses

We will do a sensitivity analysis to test whether the gap between BAS and KA would influence the obtained result by limiting the gap ≤12 months, 13-24 months and >24 months. To investigate whether the type of Bariatric Surgery (BAS), such as gastric banding or gastric bypass, has an impact on the outcomes, we plan to conduct a sensitivity analysis. This will involve narrowing our focus to each specific type of BAS. This particular approach has not been previously applied, and the findings could prove to be significant.

## Patient and Public Involvement (PPI)

This project follows the EULAR recommendations for the inclusion of patient representatives in the contemporary scientific process.<sup>46</sup> This protocol was introduced to a Danish PPI. The research questions and the reported outcomes was discussed from the PPI perspectives.

#### **HEALTH RESEARCH ETHICS AND GENERAL CONSIDERATIONS**

# **Funding**

Section for Biostatistics and Evidence-Based Research, the Parker Institute, Bispebjerg and Frederiksberg Hospital is supported by a core grant from the Oak Foundation (OCAY-18-774-OFIL). Saber M. Saber is supported by a grant from Karen Elise Jensens Fond. The supporting institutions had no role in study design or writing of this protocol.

### Conflict of interest

All will be disclosed.

#### **Disclaimers**

The views expressed in the submitted protocol are the authors' own and not an official position of the institution or funder.

### **Ethics**

In Denmark, the Act on Processing of Personal Data does not require ethical permission or obtained consent for anonymised retrospective register studies. The Danish Data Protection Agency has approved the study with nr p-2023-14433.

## **R**EFERENCES

1. Evans, J.T., et al. How long does a knee replacement last? A systematic review and meta-analysis of case series and national registry reports with more than 15 years of follow-up. The Lancet 393, 655-663 (2019).

- 2. M., K., O., G., G. & S., H.F. The epidemiology of failure in total knee arthroplasty. *The Bone & Joint Journal* **98-B**, 105-112 (2016).
- 3. Lenguerrand, E., et al. Risk factors associated with revision for prosthetic joint infection following knee replacement: an observational cohort study from England and Wales. *The Lancet Infectious Diseases* **19**, 589-600 (2019).
- 4. Jasper, L., Jones, A., Mollins, J., Pohar, S. & Beaupre, L. Risk factors for revision of total knee arthroplasty: A scoping review. *BMC Musculoskeletal Disorders* **17**(2016).
- 5. Onggo, J.R., Ang, J.J.M., Onggo, J.D., de Steiger, R. & Hau, R. Greater risk of all-cause revisions and complications for obese patients in 3 106 381 total knee arthroplasties: a meta-analysis and systematic review. *ANZ Journal of Surgery* 91, 2308-2321 (2021).
- 6. Rassir, R., Sierevelt, I.N., van Steenbergen, L.N. & Nolte, P.A. Is obesity associated with short-term revision after total knee arthroplasty? An analysis of 121,819 primary procedures from the Dutch Arthroplasty Register. *The Knee* 27, 1899-1906 (2020).
- 7. Boyce, L., *et al.* The outcomes of total knee arthroplasty in morbidly obese patients: a systematic review of the literature. *Archives of Orthopaedic and Trauma Surgery* **139**, 553-560 (2019).
- 8. Chaudhry, H., et al. Revision Rates and Functional Outcomes Among Severely, Morbidly, and Super-Obese Patients Following Primary Total Knee Arthroplasty: A Systematic Review and Meta-Analysis. *JBJS Rev* 7, e9 (2019).
- 9. O'Brien, P.E., et al. Long-Term Outcomes After Bariatric Surgery: a Systematic Review and Metaanalysis of Weight Loss at 10 or More Years for All Bariatric Procedures and a Single-Centre Review of 20-Year Outcomes After Adjustable Gastric Banding. *Obes Surg* 29, 3-14 (2019).
- 10. Estimate of Bariatric Surgery Numbers, 2011-2020, accessed 04.11.2022. Vol. 2022.
- 11. Chang, S.H., *et al.* Early major complications after bariatric surgery in the USA, 2003-2014: a systematic review and meta-analysis. *Obes Rev* **19**, 529-537 (2018).
- 12. Contival, N., Menahem, B., Gautier, T., Le Roux, Y. & Alves, A. Guiding the non-bariatric surgeon through complications of bariatric surgery. *J Visc Surg* **155**, 27-40 (2018).
- 13. Patel, J.J., Mundi, M.S., Hurt, R.T., Wolfe, B. & Martindale, R.G. Micronutrient Deficiencies After Bariatric Surgery: An Emphasis on Vitamins and Trace Minerals [Formula: see text]. *Nutr Clin Pract* **32**, 471-480 (2017).
- Li, S., et al. Does Prior Bariatric Surgery Improve Outcomes Following Total Joint Arthroplasty in the Morbidly Obese? A Meta-Analysis. *J Arthroplasty* **34**, 577-585 (2019).
- 15. Smith, T.O., T, Hing, C.B. & Macgregor, A. Does bariatric surgery prior to total hip or knee arthroplasty reduce post-operative complications and improve clinical outcomes for obese patients? *The Bone & Joint Journal* **98-B**, 1160-1166 (2016).
- 16. Dowsey, M.M., *et al.* Effect of Bariatric Surgery on Risk of Complications After Total Knee Arthroplasty. *JAMA Network Open* **5**, e226722 (2022).
- 17. McLawhorn, A.S., et al. Bariatric Surgery Improves Outcomes After Lower Extremity Arthroplasty in the Morbidly Obese: A Propensity Score-Matched Analysis of a New York Statewide Database. *J Arthroplasty* 33, 2062-2069 e2064 (2018).
- 18. Wang, Y., *et al.* Impact of Bariatric Surgery on Inpatient Complication, Cost, and Length of Stay Following Total Hip or Knee Arthroplasty. *J Arthroplasty* **34**, 2884-2889 e2884 (2019).
- 19. Liu, J.X., Paoli, A.R., Mahure, S.A., Bosco, J., 3rd & Campbell, K.A. Preoperative Bariatric Surgery and the Risk of Readmission Following Total Joint Replacement. *Orthopedics* **41**, 107-114 (2018).

20. Liu, J.X., Paoli, A.R., Mahure, S.A., Bosco, J., 3rd & Campbell, K.A. Preoperative Bariatric Surgery Utilization Is Associated With Increased 90-day Postoperative Complication Rates After Total Joint Arthroplasty. *J Am Acad Orthop Surg* 28, e206-e212 (2020).

- Ighani Arani, P., Wretenberg, P., Ottosson, J., Robertsson, O. & W-Dahl, A. Bariatric surgery prior to total knee arthroplasty is not associated with lower risk of revision: a register-based study of 441 patients. *Acta Orthopaedica* **92**, 97-101 (2021).
- R., M.J., D., W.C. & J., T.M. Bariatric surgery does not improve outcomes in patients undergoing primary total knee arthroplasty. *The Bone & Joint Journal* **97-B**, 1501-1505 (2015).
- Werner, B.C., Kurkis, G.M., Gwathmey, F.W. & Browne, J.A. Bariatric Surgery Prior to Total Knee Arthroplasty is Associated With Fewer Postoperative Complications. *The Journal of Arthroplasty* **30**, 81-85 (2015).
- Inacio, M.C.S., *et al.* Bariatric Surgery Prior to Total Joint Arthroplasty May Not Provide Dramatic Improvements in Post-Arthroplasty Surgical Outcomes. *The Journal of Arthroplasty* **29**, 1359-1364 (2014).
- 25. Mocarski, M., Tian, Y., Smolarz, B.G., McAna, J. & Crawford, A. Use of International Classification of Diseases, Ninth Revision Codes for Obesity: Trends in the United States from an Electronic Health Record-Derived Database. *Population Health Management* 21, 222-230 (2017).
- 26. Benchimol, E.I., et al. The REporting of studies Conducted using Observational Routinely-collected health Data (RECORD) statement. *PLoS Med* **12**, e1001885 (2015).
- 27. Schmidt, M., Pedersen, L. & Sørensen, H.T. The Danish Civil Registration System as a tool in epidemiology. *Eur J Epidemiol* **29**, 541-549 (2014).
- Pedersen, A.B., Mehnert, F., Odgaard, A. & Schroder, H.M. Existing data sources for clinical epidemiology: The Danish Knee Arthroplasty Register. *Clin Epidemiol* 4, 125-135 (2012).
- 29. Schelde, A.B., *et al.* Validation of registration of pharmacological treatment in the Danish Hip and Knee Arthroplasty Registers. *Basic & Clinical Pharmacology & Toxicology* **128**, 455-462 (2021).
- 30. Voldstedlund, M., Haarh, M. & Mølbak, K. The Danish Microbiology Database (MiBa) 2010 to 2013. *Euro Surveill* **19**(2014).
- 31. Schmidt, M., et al. The Danish National Patient Registry: a review of content, data quality, and research potential. *Clinical epidemiology* **7**, 449-490 (2015).
- 32. Kildemoes, H.W., Sørensen, H.T. & Hallas, J. The Danish National Prescription Registry. *Scand J Public Health* **39**, 38-41 (2011).
- 33. Baadsgaard, M. & Quitzau, J. Danish registers on personal income and transfer payments. *Scand J Public Health* **39**, 103-105 (2011).
- 34. Jensen, V.M. & Rasmussen, A.W. Danish Education Registers. Scand J Public Health 39, 91-94 (2011).
- 35. McNally, M., *et al.* The EBJIS definition of periprosthetic joint infection. *Bone Joint J* **103-b**, 18-25 (2021).
- 36. Milandt, N.R., Gundtoft, P.H. & Overgaard, S. A Single Positive Tissue Culture Increases the Risk of Rerevision of Clinically Aseptic THA: A National Register Study. *Clin Orthop Relat Res* **477**, 1372-1381 (2019).
- 37. Tande, A.J. & Patel, R. Prosthetic joint infection. *Clin Microbiol Rev* **27**, 302-345 (2014).
- Pedersen, A.B., Mehnert, F., Johnsen, S.P. & Sørensen, H.T. Risk of revision of a total hip replacement in patients with diabetes mellitus: a population-based follow up study. *J Bone Joint Surg Br* **92**, 929-934 (2010).
- Jämsen, E., et al. Obesity, diabetes, and preoperative hyperglycemia as predictors of periprosthetic joint infection: a single-center analysis of 7181 primary hip and knee replacements for osteoarthritis. J Bone Joint Surg Am 94, e101 (2012).
- 40. Simpson, P.M.S., Brew, C.J., Whitehouse, S.L., Crawford, R.W. & Donnelly, B.J. Complications of Perioperative Warfarin Therapy in Total Knee Arthroplasty. *The Journal of Arthroplasty* **29**, 320-324 (2014).

Ross, A.J., Ross, B.J., Lee, O.C., Guild, G.N., 3rd & Sherman, W.F. The Impact of Prior Fragility Fractures on Complications After Total Hip Arthroplasty: A Propensity Score-Matched Cohort Study. *Arthroplast Today* 11, 41-48 (2021).

- 42. Elixhauser, A., Steiner, C., Harris, D.R. & Coffey, R.M. Comorbidity Measures for Use with Administrative Data. *Medical Care* **36**, 8-27 (1998).
- Ondeck, N.T., et al. Discriminative Ability of Elixhauser's Comorbidity Measure is Superior to Other Comorbidity Scores for Inpatient Adverse Outcomes After Total Hip Arthroplasty. *J Arthroplasty* 33, 250-257 (2018).
- Gordon, M., Stark, A., Sköldenberg, O.G., Kärrholm, J. & Garellick, G. The influence of comorbidity scores on re-operations following primary total hip replacement. *The Bone & Joint Journal* **95-B**, 1184-1191 (2013).
- 45. Austin, P.C. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. *Multivariate Behavioral Research* **46**, 399-424 (2011).
- 46. De Wit, M.P.T., *et al.* European League Against Rheumatism recommendations for the inclusion of patient representatives in scientific projects. *Annals of the Rheumatic Diseases* **70**, 722-726 (2011).